CLINICAL TRIAL: NCT05783973
Title: A Single-Center Exploratory Study to Assess the Feasibility in Bile cfDNA of Resectable Biliary Tract Carcinomas by Using Burning Rock Gene Testing Platform
Brief Title: Study to Assess the Feasibility in Bile cfDNA of Resectable Biliary Tract Carcinomas
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2023-043-02
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-02

CONDITIONS: This Study Aims to Reveal the Effectiveness, Accuracy, and Feasibility in Bile
Keywords: resectable BTC，tissue, blood , and bile samples，genomic alterations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- bile group: bile samples from 20 resectable BTC patients with 520 Panel sequencing (bile10000X)
  Interventions: Diagnostic Test: Next generation sequencing
- Tissue group: tissue samples from 20 resectable BTC patients with 520 Panel sequencing (tissue1000X)
  Interventions: Diagnostic Test: Next generation sequencing
- Plasma group: plasma samples from 20 resectable BTC patients with 520 Panel sequencing (plasma 10000X)
  Interventions: Diagnostic Test: Next generation sequencing

INTERVENTIONS:
Diagnostic Test: Next generation sequencing — Extract DNA from bile，tissue and tissue sample, minimum DNA amount should be over 50ng.

SUMMARY:
This study intends to use Onconscreen plus 520 Panel (Burning Rock, China) to conduct NGS testing in matched tissue, blood , and bile samples of patients with Resectable Biliary Tract Carcinomas（BTC）. In order to explore thefeasibility in bile cfDNA of BTC，we will collect relevant clinical information and follow-up treatment information. This study aims to reveal the effectiveness, accuracy, and feasibility in bile, as compared to tissues and blood samples.

DETAILED DESCRIPTION:
In this study, we will investigate the potential of bile for genomic alterations using matched tissue, plasma and bile from 20 Resectable BTC Patients。The patient samples will be submitted for next-generation sequencing (NGS)，The results will include but will not be limited to genomic profling, tumor mutation burden (TMB), microsatellite instability (MSI) status, homologous recombination repair deficiency (HRD)。Patients will be followed-up for treatment responses until radiological confirmation of disease recurrence ,The molecular assay results will then be analyzed with clinical data including objective responses disease-free survival outcomes, among others, to reveal the effectiveness, accuracy, and feasibility in bile, as compared to tissues and blood samples.

Baseline tissues, plasma and sputum samples from 20 Resectable BTC Patients with 520 Panel sequencing (tissue 1000X, ,plasma cfDNA 10000X，bile 10000X), in different methods will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are diagnosed with diagnosed with BTC (including IHCC、EHCC、GBC)by histology or cytology
2. Patients who signed informed consent form;
3. Patients who agree and have the ability to follow the planned research visits, provide surgical tissue, blood, and bile samples, provide clinical information, and cooperate with other research steps.

Exclusion Criteria:

a.Patients who be deemed unsuitable for enrollment by the researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Planning to enroll 20 resectable BTC patients, age over 18 years old following the eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-02-02 (Estimated)

PRIMARY OUTCOMES:
Compare different sample types with concordence rate, sensitivity, and specificity. | 1 years
  Concordance rate was defined as the fraction of the total number of true positive and true negative patients relative to the cohort or indicated subgroup; Sensitivity rate means true positive rate, true positive patients were defined as those who carried at least one genomic alteration that were detected in both matched samples.
  Specificity rate means ture negative rate, patients were as defined true negative if no alteration was detected from either matched sample.

CONTACTS AND LOCATIONS:
Overall Officials: Changzhen Shang, MD, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided